CLINICAL TRIAL: NCT04545502
Title: A Prospective and Retrospective, Multi-Centre, Post-Market, Non-Interventional Study of Terumo Aortic Knitted and Woven Grafts, and Cardiovascular Patches
Brief Title: PANTHER Study of Terumo Aortic Knitted and Woven Grafts, and Cardiovascular Patches
Acronym: PANTHER
Status: Recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PANTHER-001
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Aneurysm; Dissection; Aortic Root Aneurysm; Aortic Root Dissection; Carotid Artery Injuries; Aortic Arch; Bypass Extremity Graft; Occlusive Vascular Disease; Aortic Diseases
Keywords: Vascular Surgery
MeSH Terms: conditions — Aneurysm; Aortic Root Aneurysm; Dissection, Ascending Aorta; Carotid Artery Injuries; Aortic Diseases | interventions — Vascular Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Gelsoft Plus - Straights and Bifurcated: Patients with aneurysmal or occlusive disease, including those with connective tissue disorders who have received/will receive a Gelsoft Plus Straight or Bifurcate, implanted in the abdomen or peripheral arteries in the last 5 years and from study launch onwards.
  Interventions: Device: Gelsoft Plus Vascular Graft
- Gelsoft Plus - Extra-Anatomical: Any patients who have received/will receive a Gelsoft Plus Extra-Anatomical supported or unsupported graft, implanted for: axillary-femoral bypass, femoral-femoral bypass or femoral-popliteal bypass in the last 5 years and from study launch onwards.
  Interventions: Device: Vascular Bypass Graft
- Cardiovascular Patches - Gelseal, Gelsoft, Thin Wall: Patients who have been implanted with/require a cardiovascular patch for: thoracic vessel repair with a Gelseal Cardiovascular Patch; abdominal or peripheral vessel repair with a Gelsoft Cardiovascular Patch; or carotid endarterectomy with a Thin Wall Carotid Patch in the last 5 years and from study launch onwards.
  Interventions: Device: Cardiovascular Patch
- Gelweave - Abdominal, Thoracic, Thoracoabdominal: Patients who, due to either aneurysmal or occlusive disease, have had/require vascular repair of one of the following, implanted in the last 5 years and from study launch onwards:
  * Abdominal aorta, arteries arising from the abdominal aorta or peripheral arteries including femoral, iliac and popliteal arteries.
  * Thoracic aorta or arteries arising from the thoracic aorta.
  * Abdominal and thoracic aorta requiring a thoracoabdominal repair
  Interventions: Device: Gelweave Vascular Graft
- Gelweave - Valsalva: Patients who have had/require aortic root repair using valve sparing or valve replacing procedures, with or without replacement of the aortic arch, implanted in the last 5 years and from study launch onwards.
  Interventions: Device: Gelweave Valsalva Vascular Graft

INTERVENTIONS:
Device: Gelsoft Plus Vascular Graft — Gelatin coated, knitted vascular prosthesis implanted to act as a conduit for channeling blood during repair of damaged or diseased vessels.
  Other Names: Gelsoft Plus
  Groups: Gelsoft Plus - Straights and Bifurcated
Device: Vascular Bypass Graft — Gelatin coated, knitted vascular prosthesis implanted to act as an extra-anatomical bypass for channeling blood during repair of damaged or diseased vessels.
  Other Names: Gelsoft Plus Extra Anatomical
  Groups: Gelsoft Plus - Extra-Anatomical
Device: Cardiovascular Patch — Cardiovascular knitted polyester patches are frequently used to treat the carotid or femoral arteries to prevent stroke and repair damage to vessels.
  Other Names: Gelseal Patch; Gelsoft Patch; Thinwall Patch; Cardiovascular Fabrics
  Groups: Cardiovascular Patches - Gelseal, Gelsoft, Thin Wall
Device: Gelweave Vascular Graft — The Gelweave woven polyester vascular graft allows replacement of large sections of arteries and, following anastomosis to the native blood vessel, provides a stable conduit for blood flow.
  Other Names: Gelweave
  Groups: Gelweave - Abdominal, Thoracic, Thoracoabdominal
Device: Gelweave Valsalva Vascular Graft — This woven polyester graft is designed to match the aortic root anatomy and is implanted to repair or replace a portion of the aorta in case of an aneurysm, dissection or coarctation at the level of the thoracic aorta.
  Other Names: Gelweave Valsalva
  Groups: Gelweave - Valsalva

SUMMARY:
The purpose of this registry is to collect safety and performance data on all commercially available Terumo Aortic knitted and woven grafts, and cardiovascular patches in standard clinical practice.

Data will be collected both retrospectively and prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria in order to be eligible for inclusion in the study:

All Patients:

* Patient meets the minimum age as per local regulations at time of consent
* Patient requires treatment with study device(s) according to the IFU(s)
* Patient is willing and able to comply with all SOC procedures and study visits
* Patient or their legally authorised representative (LAR) has given written informed consent to participate in study, including consent to collect data retrospectively

  * For prospective emergency patients, retrospective consent is permissible
  * For retrospective patients who are deceased at time of enrollment, local EC regulations relating to consent process should be followed.

Retrospective Patients only:

* Patient has a minimum of 1 year post-operative follow-up data available, or complete data to death.
* Patient implant date is no more than 5 years prior to study start date.

Exclusion Criteria:

* Any patient who meets any of the following exclusion criteria will be excluded from participation in the study:

  * Patient is unable or unwilling to comply with the SOC procedures or follow-up regime
  * Patient is contraindicated per the device IFU
  * Patient has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre- and post-procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require treatment, or have already received treatment within the last 5 years, with the following commercially available Terumo Aortic knitted and woven grafts and cardiovascular patches:
  * Gelsoft Plus - Straights and Bifurcated
  * Gelsoft Plus - Extra-Anatomical
  * Cardiovascular Patches - Gelseal, Gelsoft and Thin Wall
  * Gelweave - Abdominal, Thoracic and Thoracoabdominal
  * Gelweave - Valsalva This is a non-interventional study and therefore only patients who would normally receive treatment with a Terumo Aortic devices as part of standard treatment at the participating institution can be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2037-01 (Estimated)

PRIMARY OUTCOMES:
Operative Death | 1 Year
  30 Day or In-Hospital Mortality
Graft Leakage | 1 Year
  Device Failure: The presence of leakage or excessive bleeding through graft/patch

SECONDARY OUTCOMES:
Device Endpoints | 1 Year
  Device failures, requirement for reintervention or device related adverse events
Procedural Endpoints | 1 Year
  Rifampicin or heparin soaking, procedure related adverse events
Safety Endpoints | 1 Year
  Occurrence of the following: Mortality, Ischemia, Occlusion, Thrombosis, Haemmorrhage, Rupture, Pseudoaneurysm, Stroke

CONTACTS AND LOCATIONS:
Locations (31):
- United States (10):
  - University of Colorado Anschutz, Aurora, Colorado
  - University of South Florida - Tampa General, Tampa, Florida
  - Indiana University Health, Indianapolis, Indiana
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Belgium (3):
  - UZ Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
- Hamilton General, Hamilton, Ontario, Canada
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Lille, Lille
  - Hôpital Nord Marseille, Marseille
  - CHU de Rennes, Rennes
  - Hôpitaux Universitaires de Strasbourg - Hôpital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
- Germany (7):
  - Charité Berlin, Berlin
  - Uniklinik Bonn, Bonn
  - UNIVERSITÄTSKLINIKUM FREIBURG/Bad Krozingen, Freiburg im Breisgau
  - UKE Hamburg, Hamburg
  - Heart Center Leipzig, Leipzig
  - Universitätsmedizin Mainz (University Hospital Mainz), Mainz
  - Ludwig-Maximilian Universität (LMU) Klinikum, Munich
- Semmelweis University Heart and Vascular Center, Budapest, Budapest, Hungary
- Amphia Hospital (Ziekenhuis) Breda, Breda, Netherlands